CLINICAL TRIAL: NCT01721382
Title: Treatment of Dysglycemia Using Sitagliptin in Adolescents With Cystic Fibrosis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Larry Fox, Pediatric Endocrinologist, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CFRD-01
Record Dates: First submitted 2012-10-26; First posted 2012-11-05 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; CF; CFRD; sitagliptin; incretins; GLP1; GIP; beta cell function; adolescents
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sitagliptin (Experimental): Treatment with sitagliptin
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin

SUMMARY:
This pilot study will be conducted in adolescents with cystic fibrosis (CF) without diabetes but with abnormal glucose tolerance, and will assess the effects of sitagliptin on glucose regulation. An oral glucose tolerance test (OGTT) and a mixed meal tolerance test (MMTT), will be performed at baseline and again ~4 weeks after treatment with study drug. We will also look at blood sugars throughout the day using a continuous glucose monitor (CGM) before each time the MMTT/OGTT are performed. Several hormones that may affect the way the body regulates blood sugars will be measured in blood when the OGTT and MMTT are done. We will assess the effect this medicine has on blood sugars (using CGM) and the effect the medicine has on the hormones measured during the OGTT and MMTT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF between 13 and <21 yrs old
* Known impaired or indeterminate glucose tolerance (based on a prior OGTT)
* No history of CFRD

Exclusion Criteria:

* Insulin use in the last two months
* Acute pulmonary exacerbation / oral corticosteroid use in the last 6 weeks
* History of pancreatitis in the last 12 months
* Skin rashes or conditions that may affect CGM placement and wear
* Pregnancy or intent on becoming pregnant
* Patients on growth hormone therapy
* Renal insufficiency with creatinine clearance <50 ml/min (based on Schwartz formula)

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Response to sitagliptin | Change from baseline to ~4 weeks of study drug
  Baseline and stimulated C-peptide levels (using mixed meal tolerance test) before and after treatment with sitagliptin.
Response to sitagliptin | Change from baseline to ~4 weeks of study drug
  Change in glycemic variability using continuous glucose monitoring data before and after treatment with dipeptidyl peptidase-4 inhibitor.
Response to sitagliptin | Change from baseline to ~4 weeks of study drug
  Change in incretins concentrations (glucagon like peptide 1; glucose-dependent insulinotropic polypeptide) in response to study drug.
Response to sitagliptin | Change from baseline to ~4 weeks of study drug
  Change in incretin (glucagon like peptide 1; glucose-dependent insulinotropic polypeptide) concentrations in response to study drug.

SECONDARY OUTCOMES:
Beta-cell function | Change from baseline to ~4 weeks of study drug
  Beta-cell function will be measured using mixed meal tolerance tests (MMTT) and oral glucose tolerance tests (OGTT), assessing maximum concentration and area under the curve (AUC) of glucose, insulin and c-peptide for both OGTT and MMTT.
Continuous glucose monitoring (CGM) | change from baseline to ~4 weeks of study drug
  Baseline and post-treatment changes in glycemic variability using CGM, including mean amplitude of glycemic excursion (MAGE), peak post-prandial blood sugars, and glucose area under the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Fox, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States